CLINICAL TRIAL: NCT04177186
Title: Effectiveness of Strength Training After Administration of Botulinum Toxin in Children With Spastic Diplegic and Hemiplegic Cerebral Palsy on Muscle Volume and Gross Motor Function: A Prospective, Double-blind, Randomized Clinical Trial
Brief Title: Strength Training in Children With Spastic Diplegic and Hemiplegic Cerebral Palsy Receiving Botulinum Toxin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Associate professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MMDU/2019/03; U1111-1240-0890 (Other: UTN by WHO international clinical Trial Registry Platform)
Record Dates: First submitted 2019-11-20; First posted 2019-11-26 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Spastic Diplegic Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: Cerebral palsy; Botox
MeSH Terms: conditions — Cerebral Palsy | interventions — Resistance Training; Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will follow double-blinding/ masking. As the outcome assessor and the participant will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strength training group (Experimental): ST group only strength training will be provided.
  Interventions: Other: Strength training
- strength training with botulinum toxin (Experimental): BT-ST group, strength training will be provided after the administering Botulinum toxin into the muscle belly guided under Ultra sound imaging.
  Interventions: Combination Product: Strength training with botulinum toxin

INTERVENTIONS:
Other: Strength training — Strength training for hamstring and gastrocnemius only, pre and post 12 weeks of intervention
  Arms: strength training group
Combination Product: Strength training with botulinum toxin — Strength training for hamstring and gastrocnemius with Ultra Sound Imaging method, pre and post 12 weeks of intervention
  Arms: strength training with botulinum toxin

SUMMARY:
To estimate the effectiveness of strength training after administration of botulinum toxin in children with spastic diplegic cerebral palsy and hemiplegic cerebral palsy on muscle volume and gross motor function. Forty Children with spastic diplegic cerebral palsy (CSDP) and children with hemiplegic cerebral palsy (CHCP) in GMFCS levels I, II and III will be recruited by the convenience sampling method. Thickness of both hamstring and gastrocnemius will be recorded with Ultra Sound Imaging method, pre and post 12 weeks of intervention. In ST group only strength training will be provided. While in BT-ST group, strength training will be provided after the administering Botulinum toxin into the muscle belly guided under Ultra sound imaging. Pre-post intervention differences in muscle thickness and gross motor function will be recorded and analysed.

DETAILED DESCRIPTION:
Botulinum toxin is a neurotransmitter produced by clostridium Botulinum. It is the one of the most beneficial method for treating spasticity and providing functional improvement. By reducing the spasticity, the available muscle can be utilized to perform functional activities. Muscle volume decreases following the administration of Botulinum toxin to the neuromuscular junction. Strength training has positive impact on improving muscle volume. There are few studies are available regarding the exercise training following the administration of Botulinum toxin to the neuromuscular junction. But to the best of the investigators knowledge, there is no study available regarding the effectiveness of strength training on muscle volume and gross motor function following the administration of Botulinum toxin to the neuromuscular junction.2. To determine the effectiveness of strength training on muscle volume estimated by Ultrasound imaging following the administration of Botulinum toxin to hamstring and gastrocnemius is the objective of the study. The study protocol was approved by the institutional research advisory committee (RAC) and registered under the Universal Trial Number (UTN), U1111-1240-0890. The protocol will be registered under ClinicalTrials.gov, under World Health Organization International Clinical Trials Registry Platform and then the study will be submitted for the ethical approval by institutional ethics committee of Maharishi Markandeshwar Deemed to Be University, Mullana, and Haryana with unique reference number. The study will be executed in accordance with the principles of the Declaration of Helsinki (Revised, 2013) and National ethical guidelines for Biomedical and Health research involving human participants by Indian council for medical research (ICMR, 2017). The purpose of the study will be clearly explained to the patient with Head and neck cancer. Written informed consent form will be obtained from the recruited patients. Total of X CSDCP and CHCP will be screened and through convenience sampling method, 34 children will be selected based on the inclusion criteria for the cross-over trail design. Demographic data will be recorded for all the recruited children.

.

ELIGIBILITY:
Inclusion Criteria:

* Children with spastic diplegic cerebral palsy (CSDP) and children with hemiplegic cerebral palsy (CHCP) in GMFCS level I, II and III.
* CSDCP and CHCP aged between 5 to 17 years
* Ankle dorsiflexion <5°
* Knee extension < 90°

Exclusion Criteria:

* CSDCP and CHCP with any type of lower limb surgery within 3 months
* Children who are not willing to participate in the study

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-11-18 (Estimated)

PRIMARY OUTCOMES:
Ultra-Sound imaging | Change from baseline, and post 12 weeks of intervention will be measured.
  Muscle thickness measured through Ultra-Sound imaging
Gross motor function measure- 88 | Change from baseline, and post 12 weeks of intervention will be measured.
  Gross motor function measure- 88 helps in measuring the activities in standing and walking.

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, MPT, Principal Investigator — Maharishi Markandeshwar institute of Physiotherapy and Rehabilitation, Mullana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yigitoglu P, Kozanoglu E. Effectiveness of electrical stimulation after administration of botulinum toxin in children with spastic diplegic cerebral palsy: A prospective, randomized clinical study. Turk J Phys Med Rehabil. 2019 Feb 4;65(1):16-23. doi: 10.5606/tftrd.2019.2236. eCollection 2019 Mar. PMID 31453540
- [Background] Juneja M, Jain R, Gautam A, Khanna R, Narang K. Effect of multilevel lower-limb botulinum injections & intensive physical therapy on children with cerebral palsy. Indian J Med Res. 2017 Nov;146(Supplement):S8-S14. doi: 10.4103/ijmr.IJMR_1223_15. PMID 29578189
- [Background] Williams SA, Reid S, Elliott C, Shipman P, Valentine J. Muscle volume alterations in spastic muscles immediately following botulinum toxin type-A treatment in children with cerebral palsy. Dev Med Child Neurol. 2013 Sep;55(9):813-20. doi: 10.1111/dmcn.12200. Epub 2013 Jun 22. PMID 23789782
- [Background] Hastings-Ison T, Blackburn C, Rawicki B, Fahey M, Simpson P, Baker R, Graham K. Injection frequency of botulinum toxin A for spastic equinus: a randomized clinical trial. Dev Med Child Neurol. 2016 Jul;58(7):750-7. doi: 10.1111/dmcn.12962. Epub 2015 Nov 20. PMID 26589633
- [Background] Kaushik PS, Gowda VK, Shivappa SK, Mannapur R, Jaysheel A. A Randomized Control Trial of Botulinum Toxin A Administration under Ultrasound Guidance against Manual Palpation in Spastic Cerebral Palsy. J Pediatr Neurosci. 2018 Oct-Dec;13(4):443-447. doi: 10.4103/JPN.JPN_60_18. PMID 30937086
- See also: A Randomized Control Trial of Botulinum Toxin A Administration under Ultrasound Guidance against Manual Palpation in Spastic Cerebral Palsy. — https://www.ncbi.nlm.nih.gov/pubmed/30937086